CLINICAL TRIAL: NCT04634825
Title: A Phase 2 Open-Label Trial to Evaluate Enoblituzumab in Combination With Retifanlimab or Tebotelimab in the First-Line Treatment of Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Enoblituzumab Plus Retifanlimab or Tebotelimab in Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on internal review of safety data
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGA271-06
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Enrollment into each cohort will occur independently in a non-randomized fashion, based on PD-L1 expression results. Patients may not crossover between cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Retifanlimab Cohort (Experimental): Enoblituzumab 15 mg/kg every 3 weeks plus retifanlimab 375 mg every 3 weeks for up to 35 cycles
  Interventions: Biological: Enoblituzumab; Biological: Retifanlimab
- Tebotelimab Cohort (Experimental): Enoblituzumab 15 mg/kg every 3 weeks plus tebotelimab 600 mg every 3 weeks for up to 35 cycles
  Interventions: Biological: Enoblituzumab; Biological: Tebotelimab

INTERVENTIONS:
Biological: Enoblituzumab — Anti-B7-H3 antibody
  Other Names: MGA271
Biological: Retifanlimab — Anti-PD-1 antibody
  Other Names: INCMGA00012; MGA012; Zynyz
  Arms: Retifanlimab Cohort
Biological: Tebotelimab — PD-1 X LAG-3 bispecific DART molecule
  Other Names: MGD013
  Arms: Tebotelimab Cohort

SUMMARY:
This is a Phase 2 study of enoblituzumab combined with either retifanlimab or tebotelimab administered as first-line treatment to patients with recurrent or metastatic squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) not curable by local therapy
* No prior systemic therapy for SCCHN in the recurrent or metastatic setting (with the exception of systemic therapy completed > 6 months prior if given as part of multimodal treatment for locally advanced disease)
* Primary tumor locations of oropharynx, oral cavity, hypopharynx, or larynx. Patients may not have a primary tumor site of upper esophagus, salivary gland, or nasopharynx (any histology)
* Availability of formalin-fixed, paraffin embedded tumor specimen or contemporary biopsy for immunohistochemical evaluation of pharmacodynamic markers of interest
* Willing to consent for baseline and on-treatment biopsy.
* Performance status 0 or 1
* Life expectancy of 6 months or more
* Adequate end organ function
* At least one radiographically measurable lesion
* PD-L1 expression level that is either

  1. Positive (combined positive score [CPS] ≥ 1) for the retifanlimab cohort, or
  2. Negative (CPS < 1) for the tebotelimab cohort
* Results available from human papilloma virus p16 status for oropharyngeal cancer
* Acceptable laboratory results

Exclusion Criteria:

* Disease suitable for local therapy administered with curative intent
* Progressive disease within 6 months of completion of curatively intended systemic treatment for locoregionally advanced SCCHN
* Radiation or other non-systemic therapy within 2 weeks prior to the first dose of study drug
* Prior therapy with an anti-B7-H3, anti-PD-1, anti-PD-L1, or anti-LAG-3 agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley L. Ward, MD, Study Director — MacroGenics
Locations (42):
- United States (6):
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - University of North Carolina - Lineberger Cancer Center, Chapel Hill, North Carolina
  - University of Pennsylvania - Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center- Hillman Cancer Center, Pittsburgh, Pennsylvania
- Australia (7):
  - Liverpool Hospital, Liverpool, New South Wales
  - Monash Health, Medical Oncology Department, Ruse, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Icon Cancer Centre Southport, Southport, Queensland
  - Andrew Love Cancer Centre, Barwon Health, Geelong, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Bulgaria (7):
  - Complex Oncology Center Ruse Ltd., Dobrich
  - MHAT Serdica, Panagyurishte
  - MBAL Uni Hospital, Pleven
  - MHAT Nadezhda, Medical Oncology, Sofia
  - UMHAT Tsarisa Yoanna - ISUL, Sofia
  - UMHAT Georgi Stranski Medical Oncology Department, Sofia
  - COC Dobrich, Sofia
- Hungary (5):
  - Bajcsy-Zsilinszky Korhaz, Budapest
  - Uzsoki Street Hospital, Budapest
  - Dept of Oncology, University of Debrecen, Debrecen
  - Dept of Oncology, Bekec County Hosp, Gyula
  - Dept of Oncology, Tolna County Hospital, Szekszárd
- Poland (5):
  - The Ewa Pilecka Department of Clinical Oncology, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - I Clinics of Radiotherapy and Chemiotherapy; The Maria Sklodowska-Curie National Research Institute of Oncology, Gliwice
  - Biokinetica, Józefów
  - Clinics of Head and Neck Cancer, The Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- Spain (6):
  - Complejo Hospitalario Universitario de Badajoz, Badajoz
  - Hospital Universitario Vall D'Hebrón, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Virgen de la Macarena, Seville
- Ukraine (6):
  - Communal Non-profit Enterprise "City Clinical Hospital#4" of Dnipro City, Dnipro
  - Communal Non-Profit Enterprise "Regional Center of Oncology", Oncosurgical Department of Head and Neck, Kharkiv
  - Communal Non-profit Enterprise "Regional Clinical Oncology Center of Kirovohrad Regional Council",, Kropyvnytskyi
  - Kyiv City Clinical Oncological Centre, Kyiv
  - Municipal Non-Profit Enterprise of Sumy Regional Council "Sumy Regional Clinical Oncology Dispensary", Sumy
  - Communal Nonprofit Enterprise Podilsky Regional Center of Oncology, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retifanlimab Cohort | Tebotelimab Cohort
Started | 48 | 14
Completed | 0 | 0
Not Completed | 48 | 14
Not completed — Death | 10 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study terminated by sponsor | 35 | 11
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Retifanlimab Cohort: Enoblituzumab 15 mg/kg every 3 weeks plus retifanlimab 375 mg every 3 weeks
- Tebotelimab Cohort: Enoblituzumab 15 mg/kg every 3 weeks plus tebotelimab 600 mg every 3 weeks
- Total: Total of all reporting groups
Arm/Group | Retifanlimab Cohort | Tebotelimab Cohort | Total
Number analyzed (Participants) | 48 | 14 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (11.31) | 65.1 (6.80) | 62.0 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 38 | 11 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 47 | 12 | 59
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 42 | 14 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 3 | 1 | 4
  United States | 12 | 1 | 13
  Ukraine | 12 | 2 | 14
  Poland | 6 | 1 | 7
  Bulgaria | 0 | 2 | 2
  Australia | 6 | 1 | 7
  Spain | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of Enoblituzumab Plus Retifanlimab
Description: Investigator-assessed ORR. defined as the percentage of patients in the response evaluable population who achieve the best overall response of complete response (CR) or partial response (PR),per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 criteria..
  CR is defined as disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease from baseline in the sum of diameters of target lesions
Time Frame: Tumor assessment is conducted 6 weeks after the first dose, then every 9 weeks until disease progression, up to 16.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Retifanlimab Cohort
Number analyzed (Participants) | 48
Participants | 3

2. Primary Outcome: Number of Patients With Adverse Events (AEs) Receiving Enoblituzumab Plus Tebotelimab
Time Frame: Throughout the study, up to 16.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Tebotelimab Cohort
Number analyzed (Participants) | 14
Participants | 12

3. Primary Outcome: ORR of Enoblituzumab Plus Tebotelimab
Description: Investigator-assessed ORR. ORR, defined as the percentage of patients in the response evaluable population who achieve the a best overall response of complete response (CR) or partial response (PR), per RECIST, version 1.1 criteria.
  CR is defined as disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease from baseline in the sum of diameters of target lesions
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tebotelimab Cohort
Number analyzed (Participants) | 14
Participants | 2

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from the first dose date to the date of first documented progression or death from any cause, whichever occurs first, evaluated by cohort
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Retifanlimab Cohort | Tebotelimab Cohort
Number analyzed (Participants) | 48 | 14
months | NA [NA to NA] — There was an insufficient number of events to calculate PFS. | NA [NA to NA] — There was an insufficient number of events to calculate PFS.

5. Secondary Outcome: Disease-control Rate (DCR)
Description: Percentage of response-evaluable patients with CR, PR, or stable disease (SD) for at least 3 months, evaluated by cohort
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Retifanlimab Cohort | Tebotelimab Cohort
Number analyzed (Participants) | 48 | 14
Participants | 19 | 5

6. Secondary Outcome: Duration of Response
Description: Time from the date of initial response (CR or PR) to the date of first documented progression or death from any cause, whichever occurs first, evaluated by cohort
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Retifanlimab Cohort | Tebotelimab Cohort
Number analyzed (Participants) | 48 | 14
months | NA (NA) — There were an insufficient number of progression events in the analysis population to calculate duration of response. | NA (NA) — There were an insufficient number of progression events in the analysis population to calculate duration of response.

7. Secondary Outcome: Overall Survival
Description: Time from the first dose date to the date of death from any cause, evaluated by cohort
Time Frame: up to 16.5 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Retifanlimab Cohort | Tebotelimab Cohort
Number analyzed (Participants) | 48 | 14
months | NA [NA to NA] — There were an insufficient number of death events in the analysis population to calculate overall survival. | NA [NA to NA] — There were an insufficient number of death events in the analysis population to calculate overall survival.

8. Secondary Outcome: Best Overall Response (BOR)
Description: The participants best response to treatment during their study participation. Responses are categorized as CR, PR, stable disease (SD), progressive disease (PD), or not evaluated (NE), per RECIST 1.1 criteria CR is defined as disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease from baseline in the sum of diameters of target lesions, and non-PD in non-target lesions PD is defined as at least a 20% increase from nadir in the sum of diameters of target lesions or unequivocal progression in non-target lesions SD is defined as non-PD in target and non-target lesions
Time Frame: Tumor assessment is conducted 6 weeks after first dose, then every 9 weeks until disease progression, up to 16.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Retifanlimab Cohort | Tebotelimab Cohort
Number analyzed (Participants) | 48 | 14
Participants
  Complete Response | 0 | 0
  Partial Response | 3 | 2
  Stable Disease | 20 | 5
  Progressive Disease | 15 | 2
  Not Evaluable | 10 | 5

9. Secondary Outcome: Number of Patients With AEs Receiving Enoblituzumab Plus Retifanlimab
Time Frame: Throughout the study, up to 16.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Retifanlimab Cohort
Number analyzed (Participants) | 48
Participants | 40

10. Secondary Outcome: Maximum Drug Concentration or Drug Concentration of Enoblituzumab at the End of Infusion of Enoblituzumab (Cmax)
Description: The highest measured concentration of enoblituzumab in the bloodstream.
Time Frame: Cycle 1 Day 1: Pre-infusion, end of infusion (EOI [2 hours]), 4 hours after EOI; Cycle 1 Days 2, 3, 8 and 15 at any time; On Day 1 of Cycles 2, 3, 4, 5 and 6: Pre-infusion and EOI (each cycle is 21 days)
Population: Participants who received Enoblituzumab and had at least 1 end of infusion PK sample. As pre-specified in the PK analysis plan, Enoblituzumab PK data from both arms of the study were combined for analysis since Enoblituzumab dose was schedule were consistent across both arms.
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Enoblituzumab: Enoblituzumab 15 mg/kg every 3 weeks
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 62
mcg/mL | 505.3 (130.5)

11. Secondary Outcome: Maximum Drug Concentration or Drug Concentration of Tebotelimab at the End of Infusion of Tebotelimab (Cmax)
Description: The highest measured concentration of tebotelimab in the bloodstream.
Time Frame: Cycle 1 Day 1: Pre-infusion, end of infusion (EOI [1 hour]), 4 hours after EOI; Cycle 1 Days 2, 3, 8 and 15 at any time; On Day 1 of Cycles 2, 3, 4, 5 and 6: Pre-infusion and EOI (each cycle is 21 days)
Population: Participants who received tebotelimab and had at least 1 End of Infusion PK sample
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Tebotelimab Cohort
Number analyzed (Participants) | 14
mcg/mL | 196.5 (74.8)

12. Secondary Outcome: Maximum Drug Concentration or Drug Concentration of Retifanlimab at the End of Infusion of Enoblituzumab (Cmax)
Description: The highest measured concentration of retifanlimab in the bloodstream.
Time Frame: as for outcome 11
Population: Participants who received retifanlimab and had at least 1 end of infusion PK sample.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Retifanlimab Cohort
Number analyzed (Participants) | 47
mcg/mL | 113.1 (26.9)

13. Secondary Outcome: Trough Concentration of Enoblituzumab (Ctrough or Cmin)
Description: The amount of enoblituzumab left in the bloodstream before the next dose is given.
Time Frame: Cycle 1 Day 1: Pre-infusion, end of infusion (EOI [2 hours]), 4 hours after EOI; Cycle 1 Days 2, 3, 8 and 15 at any time; On Day 1 of Cycles 2, 3, 4, 5 and 6: Pre-infusion and EOI (each cycle is 21 days
Population: Participants who received enoblituzumab and had at least 1 pre-infusion PK sample. As pre-specified in the PK analysis plan, enoblituzumab PK data from both arms of the study were combined for analysis since enoblituzumab dose and schedule were consistent across both arms.
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Enoblituzumab: Enoblituzumab 15 mg/kg
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 62
mcg/mL | 165.7 (88.8)

14. Secondary Outcome: Trough Concentration of Tebotelimab (Ctrough or Cmin)
Description: The amount of tebotelimab left in the bloodstream before the next dose is given.
Time Frame: as for outcome 11
Population: Participants who received tebotelimab and had at least 1 pre-infusion PK sample.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Tebotelimab Cohort
Number analyzed (Participants) | 12
mcg/mL | 20.1 (6.1)

15. Secondary Outcome: Trough Concentration of Retifanlimab (Ctrough or Cmin)
Description: The amount of retifanlimab left in the bloodstream before the next dose is given.
Time Frame: as for outcome 11
Population: Participants who received retifanlimab and had at least 1 pre-infusion PK sample.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Retifanlimab Cohort
Number analyzed (Participants) | 33
mcg/mL | 31.2 (15.5)

16. Secondary Outcome: Number of Patients Who Develop Antidrug Antibodies (ADA) to Enoblituzumab.
Time Frame: Prior to treatment (baseline) and at the beginning of every 3-week cycle of treatment (post baseline) up to 16.5 months
Population: As pre-specified in the PK analysis plan, enoblituzumab ADA data from both arms of the study were combined for analysis since enoblituzumab dose and schedule were consistent across both arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Enoblituzumab
Number analyzed (Participants) | 62
Participants
  Not done at baseline, negative post baseline | 3
  Not done at baseline, positive at least once post baseline | 1
  negative at baseline, not done post baseline | 6
  negative at baseline, negative post baseline | 37
  negative at baseline, positive at least once post baseline | 5
  positive at baseline, not done post baseline | 4
  positive at baseline, negative post baseline | 4
  positive at baseline, positive at least once post baseline | 2

17. Secondary Outcome: Number of Patients Who Develop ADA to Tebotelimab
Time Frame: Prior to treatment (baseline) and at the beginning of every 3-week cycle of treatment (post baseline) up to 16.5 months
Population: Only participants receiving tebotelimab were analyzed for the presence of tebotelimab ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Tebotelimab Cohort
Number analyzed (Participants) | 14
Participants
  not done at baseline, positive at least once post baseline | 1
  negative at baseline, not done post baseline | 2
  negative at baseline, negative post baseline | 7
  negative at baseline, positive at least once post baseline | 3
  positive at baseline, negative post baseline | 1

18. Secondary Outcome: Number of Patients Who ADA to Retifanlimab
Time Frame: Prior to treatment (baseline) and at the beginning of every 3-week cycle of treatment (post baseline) up to 16.5 months
Population: Only participants receiving retifanlimab were analyzed for the presence of retifanlimab ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Retifanlimab Cohort
Number analyzed (Participants) | 48
Participants
  Not done at baseline, negative post baseline | 3
  negative at baseline, not done post baseline | 8
  negative at baseline, negative post baseline | 37

ADVERSE EVENTS:
Time Frame: Throughout the study, up to 16.5 months
Description: AEs are based on physical exam, participant reports and significant abnormal laboratory values.
  AEs were not collected during the survival follow up. Serious AEs (SAEs) were collected in survival follow up, if considered related to study treatment by the investigator..
  Progression of cancer causing hospitalization or death is not considered an SAE, unless considered drug-related by the investigator.
Arm/Group | Retifanlimab Cohort | Tebotelimab Cohort
All-Cause Mortality (participants affected / at risk) | 10/48 | 3/14
Serious Adverse Events (participants affected / at risk) | 14/48 | 6/14
Other Adverse Events (participants affected / at risk) | 40/48 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retifanlimab Cohort (N=48) | Tebotelimab Cohort (N=14)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiotoxicity (Cardiac disorders) | 1 | 0
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 1
Immune-mediated endocrinopathy (Endocrine disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Cytomegalovirus gastritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fungating wound (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrostomy (Surgical and medical procedures) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retifanlimab Cohort (N=48) | Tebotelimab Cohort (N=14)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 6 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 6 | 1
Oedema peripheral (General disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 1
Asthenia (General disorders) | 0 | 2
Axillary pain (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Inadequate analgesia (General disorders) | 1 | 0
Swelling face (General disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 3 | 1
Oral candidiasis (Infections and infestations) | 3 | 0
Breakthrough COVID-19 (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Coronavirus infection (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Gastroenteritis staphylococcal (Infections and infestations) | 0 | 1
Gingival abscess (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Tracheostomy infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 4
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Incision site ulcer (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Lipase increased (Investigations) | 5 | 0
Weight decreased (Investigations) | 4 | 0
White blood cell count decreased (Investigations) | 4 | 0
Lymphocyte count decreased (Investigations) | 2 | 1
Amylase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Blood pressure increased (Investigations) | 2 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Coronavirus test positive (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 0
Embolism (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT04634825/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04634825/SAP_001.pdf